CLINICAL TRIAL: NCT01250639
Title: Type 2 Diabetes Mellitus Collaborative Genetic Study Room
Brief Title: Type 2 Diabetes Mellitus Collaborative Genetic Study on Non-aboriginal Taiwanese
Acronym: T2D2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: Academia Sinica, Taiwan (Other)
Responsible Party: Division of Metabolism and Endocrinology, Fuu-Jen Tsai
Other Study IDs: DMR99-IRB-164
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; non-aboriginal Taiwanese; Genome-wide association study
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum,urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is a cooperative project and aims to identify genetic components associated with type 2 diabetes mellitus (T2DM), which is significant for the population of non-aboriginal Taiwanese.

DETAILED DESCRIPTION:
This study is a cooperative project between Academia Sinica (AS), China Medical University Hospital (CMUH) and Chiayi Christian Hospital (CCH) and aims to identify genetic components associated with type 2 diabetes mellitus (T2DM), which is significant for the population of non-aboriginal Taiwanese. AS provides funding, designs the study protocol, and coordinates the project, including subject recruitment, collection of phenotype information and bio-specimen and quality assurance. CMUH and CCH are the study sites and are responsible for subject screening and recruitment, bio-specimen collection and packaging as well as phenotypic information collection. The study objective is to carry out a collaborative association study on T2DM in non-aboriginal Taiwanese.

A genome-wide case-control association study will be adopted. Approximately five thousand of T2DM subjects whose age is equal to or above twenty will be recruited by study physicians in the out-patient-department in CMUH and CCH. In addition, relatives of T2DM subjects with a positive family history, in which at least three family members are affected with T2DM within five generations, will be recruited by study nurses. An age-, sex-, and ethnicity-matched control will be selected randomly from the Cell Bank and Genetic Database on Non-Aboriginal Taiwanese. After obtaining informed consent, the medical history questionnaire and family background will be completed by the subjects. The subjects will be invited for a health check-up which include blood pressure, body weight, body height, waist circumference and hip circumference, as well as an ophthalmic check-up. A 15 ml of blood will be drawn from the subject for measurements of Cholesterol, HDLc, LDLc, TG, Fasting Plasma Glucose, Insulin, HbA1c, CBC without differential count, Electrolytes (Ca2+ , Na+, K+, Cl-), BUN, Creatinine, SGOT, SGPT, C-peptide, Uric Acid and CRP, as well as DNA extraction. A urine sample collection will also be requested from the subject for evaluation of urine protein, ketone body, glucose, micro albumine and creatinine.

This genome-wide association study aims to investigate the disease causing variants/genes of T2DM and diabetic subphenotypes as well as the underlying mechanisms in T2DM pathogenesis. Hopefully, early diagnostic markers and new therapies will be developed based on the genetic etiology and toward the personalized medicine in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* Subject must satisfy the diagnostic criteria for T2D at the time of examination.
* Subject is willing to participate and capable of giving informed consent.
* Subject is a self reported non-aboriginal Taiwanese, and none of the parents and grand-parents has aboriginal background.
* Relatives of T2DM subjects with a positive family history are willing to participate and capable of giving informed consent.

Exclusion Criteria:

* Type 1 Diabetes
* Gestational Diabetes
* Monogenic Diabetes
* Subject is unable to understand or give informed consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 Diabetes Mellitus
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Fuu-Jen Tsai, PHD, Principal Investigator — Division of Metabolism and Endocrinology
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan